CLINICAL TRIAL: NCT02364895
Title: ColonCancerCheck Mailed Invitations: An Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 375-2013
Record Dates: First submitted 2014-12-19; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Disorders
Keywords: Mailed invitation; Fecal Occult Blood Test; Screening

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Male arm (Experimental): Males control group: Deferred letter Males Group 1: Current CCC invitation letter Males Group 2: New letter with neutral gender content Males Group 3: New letter with male-specific content
  Interventions: Other: Males control group: Deferred letter; Other: Males Group 1: Current CCC invitation letter; Other: Males Group 2: New letter with neutral gender content; Other: Males Group 3: New letter with male-specific content
- Female arm (Experimental): Females control group: Deferred letter Females Group 1: Current CCC invitation letter Females Group 2: New letter with neutral gender content
  Interventions: Other: Females control group: Deferred letter; Other: Females Group 1: Current CCC invitation letter; Other: Females Group 2: New letter with neutral gender content

INTERVENTIONS:
Other: Males control group: Deferred letter — This letter will be sent 6 months after index (mailing) date
  Arms: Male arm
Other: Males Group 1: Current CCC invitation letter — This letter is currently used by the program in 50-54 year olds
  Arms: Male arm
Other: Males Group 2: New letter with neutral gender content — Unisex letter
  Arms: Male arm
Other: Males Group 3: New letter with male-specific content — New letter tailored for men
  Arms: Male arm
Other: Females control group: Deferred letter — This letter will be sent 6 months after index (mailing) date
  Arms: Female arm
Other: Females Group 1: Current CCC invitation letter — This letter is currently used by the program in 50-54 year olds
  Arms: Female arm
Other: Females Group 2: New letter with neutral gender content — Unisex letter
  Arms: Female arm

SUMMARY:
This study evaluates effectiveness of mailed invitations for colorectal cancer screening among screen-eligible Ontarians who are due for screening. The study will evaluate the effectiveness of mailed invitations in general (compared to no invitation) but will also determine if new invitation letters (2 letters for male, 1 letter for females) are more effective than current invitation letters used by the ColonCancerCheck program.

DETAILED DESCRIPTION:
On April 1 2008, Ontario launched Canada's first organized province-wide CRC screening program, ColonCancerCheck (CCC). CCC has a dual strategy: through the primary care physician, FOBT is offered to people aged 50 to 74 years at average risk for colorectal cancer and colonoscopy to those at increased risk based on family history. In 2010-2011, approximately 30% of Ontarians 50-74 years old were screened for colorectal cancer using the FOBT. An important factor in increasing screening participation is an invitation system.

A central tenet of organized screening programs is that all persons in the target population be invited to participate. In 2010, CCC began implementing a correspondence program in an effort to improve participation in colorectal cancer screening, starting with recall letters to individuals who were due for repeat screening two years after a normal fecal occult blood test (FOBT) and invitation letters to screen-eligible individuals who are due for screening and have not received correspondence from CCO to participate in colorectal cancer screening in the past two years to complete a screening test for colorectal cancer. Individuals who are "due for screening" includes those who have not had a FOBT in the past 2 years, a flexible sigmoidoscopy in the past 5 years, and a colonoscopy in the past 10 years. Currently, CCC sends 10,000 invitation letters monthly to 50-54 year olds only. In October 2013, the CCC correspondence program expanded to also include all eligible Ontarians 55-74 years old.

The current CCC invitation letter includes general information on the benefits of screening for colorectal cancer, the screening test itself (FOBT), and contact information to get more information. It is meant to invite individuals to speak with their primary care provider about colorectal screening. In 2013 Diego Llovet, a lead qualitative researcher at CCO, completed a series of qualitative studies examining the content of current CCC correspondence materials and made recommendations to improve the content of invitation letters. These recommendations were based on four key types of information: a) findings from seven focus groups with screen-eligible Ontarians (men and women, 50-74) who provided feedback on the messages that should be included in these letters, b) input provided by six experts in health communications and health promotion on the content and style of effective cancer screening correspondence, c) evidence from behavioral science studies on barriers to participation in colorectal cancer screening, and d) theories of health behavior change. Based on findings from focus group studies examining the content of the current CCC letter, a unisex and a male-tailored invitation letter were developed. A female-tailored letter was not developed as the focus group studies with females showed that they did not prefer female tailored messaging to a unisex one.

In the current study, we propose to test the effectiveness of mailed invitations for colorectal cancer screening in the real world setting of the CCC program. We will evaluate the effectiveness of mailed invitations in general (i.e., compared to no invitation) but we will also determine whether letters developed based on theories from behavioural science and on the results of qualitative studies with Ontarians in the target population are more effective than those currently used by the program. The findings from this study will be used to inform the CCC program correspondence but will also provide valuable information for the development of correspondence for other screening programs at Cancer Care Ontario and in other jurisdictions engaged in organized screening programs.

ELIGIBILITY:
Inclusion Criteria:

* 55-74 year old Ontarians with an active OHIP number

Exclusion Criteria:

* Death
* Withdrawn from program correspondence
* Prior colorectal cancer diagnosis
* Any FOBT activity within the last two years, including
* Flexible sigmoidoscopy within the last five years.
* Colonoscopy within the last ten years
* Other medical history in the last 30 months
* Exclusion from screening in the last 30 months
* Received a birthday letter, invitation or recall within the last two years
* Inactive primary address
* Missing address
* Address outside Ontario

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75317 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
fecal occult blood test (FOBT) uptake | 6 months after the mailing date
  Using the administrative databases at CCO, participating individuals will be followed up 6 months after the index date to measure FOBT uptake.

SECONDARY OUTCOMES:
FOBT or colonoscopy uptake | 6 months
  Using the administrative databases at CCO, participating individuals will be followed up 6 months after the index date to measure FOBT of colonoscopy uptake.
Intermediate outcomes | 8-12 weeks after mailing date
  We will mail a simple questionnaire 8-12 weeks after the index date to participants in order to assess intermediate outcomes including (a) recall of letter, (b) knowledge of colorectal cancer screening, (c) intent to be screened for colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Tinmouth, MD PhD FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre, Cancer Care Ontario

REFERENCES:
- [Derived] Tinmouth J, Llovet D, Sutradhar R, Tsiplova K, Roushani J, Lee A, Hader J, Rabeneck L, Paszat L. Two randomized controlled trials for colorectal cancer screening invitations developed using a behavioral science approach. Prev Med. 2022 Feb;155:106918. doi: 10.1016/j.ypmed.2021.106918. Epub 2021 Dec 23. PMID 34953810